CLINICAL TRIAL: NCT04665661
Title: Aerobic Exercise for Primary Dysmenorrhea: A Mixed-methods Study and Economic Evaluation
Brief Title: Aerobic Exercise for Primary Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: APD
Record Dates: First submitted 2020-11-25; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-11

CONDITIONS: Primary Dysmenorrhea
Keywords: Dysmenorrhea; Primary dysmenorrhea; Pain; Absenteeism; Academic performance
MeSH Terms: conditions — Dysmenorrhea; Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity aerobic training (HIAT) (Experimental): Women will perform treadmill-based aerobic exercise for three days a week, at 70%-85% of MHR for 30 minutes and perceived exertion of 14-16, based on the Borg RPE scale. This range39 is considered to represent HIAT. Aerobic training will be preceded by warm-up exercises for 10 minutes and followed by cool-down exercises for 10 minutes, at a perceived exertion of 11.0 (Borg RPE).
  Interventions: Behavioral: High-intensity aerobic training; Behavioral: Wait-list control
- Wait-list control (WLC) (Active Comparator): Women in the wait-list control group will be instructed to continue with their usual activities and manage their pain as normal (i.e., with analgesics).
  Interventions: Behavioral: High-intensity aerobic training; Behavioral: Wait-list control

INTERVENTIONS:
Behavioral: High-intensity aerobic training — Women will perform treadmill-based aerobic exercise for three days a week, at 70%-85% of MHR for 30 minutes and perceived exertion of 14-16, based on the Borg RPE scale. This range39 is considered to represent HIAT. Aerobic training will be preceded by warm-up exercises for 10 minutes and followed by cool-down exercises for 10 minutes, at a perceived exertion of 11.0 (Borg RPE).
Behavioral: Wait-list control — Women in the wait-list control group will be instructed to continue with their usual activities and manage their pain as normal (i.e., with analgesics).

SUMMARY:
Primary dysmenorrhea is common and can result in significant disability for many women, causing a high degree of discomfort and reduced quality of life (QoL). Our preliminary studies suggested that high-intensity aerobic training (HIAT) for 30 minutes, three times a week at 70%-85% of maximum heart rate was effective for decreasing pain and improving QoL in women suffering from primary dysmenorrhea. However, to date, no studies have evaluated the beneficial effects of HIAT on academic performance and absenteeism or the cost-effectiveness of HIAT for women with primary dysmenorrhea. Furthermore, the mechanisms underlying aerobic exercise-induced analgesia in primary dysmenorrhea remain unclear.

Here, we propose a study to address this important knowledge gap by investigating the effects of HIAT on absenteeism and academic performance among university students with primary dysmenorrhea and examine the physiological mechanisms underlying aerobic exercise-induced analgesia by conducting a fully powered, randomised, controlled crossover trial. We also propose to conduct an economic evaluation to determine the cost-effectiveness of HIAT compared with a wait-listed control group receiving usual care, according to the societal and healthcare perspectives of Hong Kong. The results of this cutting-edge research will be important for clinicians, researchers, policymakers, and women with primary dysmenorrhea. The knowledge gained from the proposed study will be useful for researchers when designing future studies to identify the mediators of pain interventions for clinical improvements, which could themselves be the target of future interventions. The findings of the proposed study will inform decision-makers regarding the extent to which existing or standard and potential interventions can improve population health (effectiveness) and the resources required to implement these interventions (costs).

DETAILED DESCRIPTION:
Objectives: (1): To evaluate the effectiveness of high-intensity aerobic training (HIAT) on pain intensity, absenteeism, and academic performance among university students with primary dysmenorrhea. (2): To investigate the physiological mechanism(s) underlying aerobic exercise-induced analgesia in women with primary dysmenorrhea. (3) Compare the cost-effectiveness of HIAT against that for usual care to treat pain associated with primary dysmenorrhea.

Design and subjects: A mixed-methods study, including a cross-over RCT, and semi-structured focus groups, alongside economic evaluation, will be conducted using 130 women with primary dysmenorrhea.

Interventions: Women will randomly allocated into high-intensity aerobic training (HIAT) or wait-list control (WLC) groups. Participants in the HIAT group will receive supervised treadmill training for the first 12 weeks of the trial. Following a four-week washout period the cross-over period will begin during Week 16, and the participants initially randomised to the WLC group will receive the HIAT regimen from Weeks 14-28. Participants initially randomized to HIAT group will be instructed not to engage in exercise during the remainder of the study period (i.e. Weeks 14-28).

Outcome measures: Pain intensity, absenteeism from university, academic performance, concentration, dysmenorrhea daily diary, and salivary progesterone and prostaglandin F2-alpha levels in saliva. The EQ-5D-3L will be used to determine the QoL for the HIAT and WLC groups.

Data analysis plan: A preliminary test using the independent samples t-test and a two-sided Student's unpaired t-test will be performed to rule out carryover effects and identify the within-participant differences in outcome variables between the study periods, respectively. Treatment effects will be evaluated using an ANOVA with a mixed-effects model considering the longitudinal repeated measures, including the effects of time within each study group and the interaction between time and intervention. The mediation effects will be assessed using the Sobel test. The EQ-5D responses will be converted into utility scores to estimate the gain or loss of quality-adjusted life-years (QUALYs). The seemingly unrelated regression (SUR) analyses will be used to estimate the total cost differences (ΔC) and effect differences (ΔE). Qualitative data will be analysed using the process of thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* women in the age group of 18-24 years old;
* non-pregnant;
* having regular menstrual cycles with cycle lengths between 24 and 30 days;
* experiencing an average menstrual pain intensity equal to or greater than 5 on a 0-10 Numerical Rating Scale; and
* scoring low (< 600 metabolic equivalent tasks [MET]/week) on the short-form of the International Physical Activity Questionnaire.

Exclusion Criteria:

* women using oral contraceptive pills, hormonal therapy, or intrauterine devices;
* women using over-the counter analgesics during menstruation to treat dysmenorrhea-associated pain and experience no pain relief with those analgesics; and
* women participating in any formal exercise programme

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity as female
Enrollment: 130 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Pre-intervention (baseline, 0 week)
  Average pain intensity during the last 24 hours during menstruation will be assessed using the 0-10 Numeric Rating Scale, with 0 representing 'No pain' and 10 representing 'Worst imaginable pain'. Higher scores indicate greater pain severity
Pain intensity | Post-intervention at 12 weeks
  Average pain intensity during the last 24 hours during menstruation will be assessed using the 0-10 Numeric Rating Scale, with 0 representing 'No pain' and 10 representing 'Worst imaginable pain'. Higher scores indicate greater pain severity
Pain intensity | Post-intervention at 28 weeks
  Average pain intensity during the last 24 hours during menstruation will be assessed using the 0-10 Numeric Rating Scale, with 0 representing 'No pain' and 10 representing 'Worst imaginable pain'. Higher scores indicate greater pain severity
Absenteeism from university | Pre-intervention (baseline, 0 week)
  A prospective electronic diary will be provided for each participant to record university absenteeism.
Absenteeism from university | Post-intervention at 12 weeks
  A prospective electronic diary will be provided for each participant to record university absenteeism.
Absenteeism from university | Post-intervention at 28 weeks
  A prospective electronic diary will be provided for each participant to record university absenteeism.
Academic performance | Pre-intervention (baseline, 0 week)
  Academic performance will be measured using the self-reported 20-item academic performance questionnaire, which was developed to measure the impacts of menstrual symptoms on academic performance. Greater scores indicate greater severity of primary dysmenorrhea
Academic performance | Post-intervention at 12 weeks
  Academic performance will be measured using the self-reported 20-item academic performance questionnaire, which was developed to measure the impacts of menstrual symptoms on academic performance. Greater scores indicate greater severity of primary dysmenorrhea
Academic performance | Post-intervention at 28 weeks
  Academic performance will be measured using the self-reported 20-item academic performance questionnaire, which was developed to measure the impacts of menstrual symptoms on academic performance. Greater scores indicate greater severity of primary dysmenorrhea
Progesterone levels | Pre-intervention (baseline, 0 week)
  Salivary levels of progesterone.
Progesterone levels | Post-intervention at 12 weeks
  Salivary levels of progesterone.
Progesterone levels | Post-intervention at 28 weeks
  Salivary levels of progesterone.
Prostaglandin F2-alpha levels | Pre-intervention (baseline, 0 week)
  Salivary levels of prostaglandin F2-alpha
Prostaglandin F2-alpha levels | Post-intervention at 12 weeks
  Salivary levels of prostaglandin F2-alpha
Prostaglandin F2-alpha levels | Post-intervention at 28 weeks
  Salivary levels of prostaglandin F2-alpha

SECONDARY OUTCOMES:
Concentration | Pre-intervention (baseline, 0 week)
  The 0-10 visual analogue scale will be used to measure the impact of dysmenorrhea on concentration, with 0 representing 'No difficulty concentrating' and 10 representing 'Maximum difficulty concentrating'.
Concentration | Post-intervention at 12 weeks
  The 0-10 visual analogue scale will be used to measure the impact of dysmenorrhea on concentration, with 0 representing 'No difficulty concentrating' and 10 representing 'Maximum difficulty concentrating'.
Concentration | Post-intervention at 28 weeks
  The 0-10 visual analogue scale will be used to measure the impact of dysmenorrhea on concentration, with 0 representing 'No difficulty concentrating' and 10 representing 'Maximum difficulty concentrating'.
Dysmenorrhea daily diary | Pre-intervention (baseline, 0 week)
  dysmenorrhea. A higher score indicates worse pain.
Dysmenorrhea daily diary | Post-intervention at 12 weeks
  The Dysmenorrhea daily diary is a questionnaire to measure the severity of dysmenorrhea. A higher score indicates worse pain.
Dysmenorrhea daily diary | Post-intervention at 28 weeks
  dysmenorrhea. A higher score indicates worse pain.
3-level version of EuroQol 5-Dimension | 12 weeks
  The 3-level version of EuroQol 5-Dimension will be used to determine the quality of life. A higher score indicates better quality of life.
Cost-diary | 12 weeks
  An electronic diary will be used to record cost expenditures in Hong Kong Dollars and work absenteeism

CONTACTS AND LOCATIONS:
Overall Officials: Priya Kannan, PhD, Principal Investigator — The Hong Kong Polytechnic Unviersity

IPD SHARING:
Plan to Share IPD: No